CLINICAL TRIAL: NCT03188809
Title: Adductor Canal Block Versus Femoral Nerve Block With Repeated Bolus Doses: Postoperative Analgesia and Functional Outcomes After Total Knee Arthroplasty
Brief Title: Adductor Canal Block Versus Femoral Nerve Block With Repeated Bolus Doses Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Seda Kurtbeyoğlu, resident, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2017-04-04; First posted 2017-06-15 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pain; Functional Outcomes
Keywords: Postoperative Pain; Functional Outcomes; Total Knee Arthroplasty; Adductor Canal Block; Femoral Nerve Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: double blind, randomised, controlled train
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- femoral nerve block (Active Comparator): Bupivacaine 0.25% will be applied to the catheter at 6 hours, when the first dose of catheter is inserted.
  Interventions: Procedure: femoral nerve block
- adductor canal block (Active Comparator): Bupivacaine 0.25% will be applied to the catheter at 6 hours, when the first dose of catheter is inserted.
  Interventions: Procedure: Adductor Canal Block

INTERVENTIONS:
Procedure: Adductor Canal Block — Adductor channel is roughly triangular in cross section and is bounded by three muscles: quadriceps anterolaterally (specifically vastusmedialis), sartorius medially and adductor magnus posteriorly. Within this canal is the femoral artery, femoral vein, the posterior branch of the obturator nerve, and branches of the femoral nerve; specifically the saphenous nerve and nerve to vastus medialis. When the femoral artery is shown by ultrasonography 21 gauge, 50 mm needle in-plane technique and the catheter will be inserted with the peripheral nerve stimulator lateral to the femoral artery. Bupivacaine 0.25% will be applied to the catheter at 6 hours, when the first dose of catheter is inserted.and the catheter will be inserted with the peripheral nerve stimulator lateral to the femoral artery. Bupivacaine 0.25% will be applied to the catheter at 6 hours, when the first dose of catheter is inserted.
  Other Names: saphen nerve block
  Arms: adductor canal block
Procedure: femoral nerve block — The probe is placed just below the inguinal crease , when the femoral artery is shown by ultrasonography, the femoral nerve stays in the lateral direction and 21 gauge, 50 mm needle will be advanced from the anterior to the posteriomedial with an in-plane technique and the catheter will be inserted by the peripheral nerve stimulator in the lateral femoral artery. Bupivacaine 0.25% will be applied to the catheter at 6 hours, when the first dose of catheter is inserted.
  Arms: femoral nerve block

SUMMARY:
After total knee prosthesis surgery, in the first postopertive days, serious pain complaints occur in the patients and this causes many problems, especially mobility limitation. For this reason, a strong analgesic is needed. As a part of multimodal analgesia after total knee surgery, nerve blocks are frequently preferred. While central nerve blocks are preferred in the forefront, peripheral nerve blocks are frequently preferred due to complications related to central nerve blocks. Femoral nerve block and adductor channel block are the preferred peripheral blocks for total knee prosthesis. Since early mobilization after total hip prosthesis is very important, it is aimed to provide sufficient analgesia by making less motor block. Previous studies have shown that adductor channel block provides similar analgesia with femoral nerve block. Early mobilization, early discharge and the impact on the risk of falls are not yet clear, although it is estimated to be in the positive direction. Again, previous studies have compared single doses and infusion doses but no repeated bolus doses. Repeated bolus doses have been shown to be more effective in studies in which adductor channel catheters have been introduced to date to compare infusion and recurrent bolus doses.

investigators aimed to compare the effects of repeated bolus doses with femoral nerve catheter and adductor channel catheter on postoperative pain and muscle strength in patients undergoing total knee replasment under spinal anesthesia in this study.

DETAILED DESCRIPTION:
After total knee prosthesis surgery, in the first postopertive days, serious pain complaints occur in the patients and this causes many problems, especially mobility limitation. For this reason, a strong analgesic is needed. As a part of multimodal analgesia after total knee surgery, nerve blocks are frequently preferred. While central nerve blocks are preferred in the forefront, peripheral nerve blocks are frequently preferred due to complications related to central nerve blocks. Femoral nerve block and adductor channel block are the preferred peripheral blocks for total knee prosthesis. Since early mobilization after total hip prosthesis is very important, it is aimed to provide sufficient analgesia by making less motor block. Previous studies have shown that adductor channel block provides similar analgesia with femoral nerve block. Early mobilization, early discharge and the impact on the risk of falls are not yet clear, although it is estimated to be in the positive direction. Again, previous studies have compared single doses and infusion doses but no repeated bolus doses. Repeated bolus doses have been shown to be more effective in studies in which adductor channel catheters have been introduced to date to compare infusion and recurrent bolus doses.

investigators aimed to compare the effects of repeated bolus doses with femoral nerve catheter and adductor channel catheter on postoperative pain and muscle strength in patients undergoing total knee revision under spinal anesthesia in this study. Materials and Methods: The patient will be informed about the procedure to be performed before the operation and written approval will be given. The patient will be premeditated with 2mg midazolam and sedayon and monitored according to routine operating room procedures and total knee prosthesis operation under spinal anesthesia. Patients will then be transferred to the collection room and ECG, NIBP and SpO2 monitoring and appropriate sterilization will be performed, and a grubby femoral nerve catheter with USG will be attached to the other group adductor channel catheter. A 20cc 0.25% marcain will be administered in 6 hours, with the first dose catheter placed in both groups.

In the compilation unit, the patient will be infused with IV PCA in the morphine. The bolus dose of 1 mg IV of the PC will be adjusted to the duration of 10 minutes of lockout. Postoperatively, 3x1 metoclopramide, 4x1 gr / 24h IV paracetamol and 3x50 mg / 24h IV dexketoprofen will be administered to each patient.

In this process, demographic information of the patients, peroperative KH, ABP, SpO2 values will be recorded. In the postoperative period, the patient's pain level, opioid requirement, motor block and muscle strength will be recorded and compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* ASA1-2-3 patients
* older than 55 years
* who undergo elective total knee prosthesis in our hospital

Exclusion Criteria:

* ASA IV patients ,
* patients with local anesthesia that we use,
* patients with coagulation disorders,
* patients with anatomical anomalies,
* patients with localized infection in the injection site ,
* patients who is incapable of using pca and/ or evaulate VAS scale,
* patients with peripheral nerve disease,
* patients with different surgical planning,
* complicated gonarthrosis patients,
* revision planned patients,
* patients who refuse to be involved in the study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative Muscle strength- Quadriceps Muscle strength scale | postoperative 48 hour
  Quadriceps Muscle strength scale

SECONDARY OUTCOMES:
postoperative analgesia - Visual analog scale | 72 hour
  Visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- SEDA, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided